CLINICAL TRIAL: NCT01958112
Title: A Single Arm, Single Stage Phase II Trial of GSK1120212 and GSK2141795 in Persistent or Recurrent Cervical Cancer
Brief Title: GSK1120212+GSK2141795 for Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-334
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cervical; Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — trametinib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSK1120212 (trametinib) and GSK2141795 (Experimental): GSK1120212 (trametinib) 1.5 mg QD + GSK2141795 50 mg QD in 28 day cycles
  Interventions: Drug: GSK1120212 (trametinib); Drug: GSK2141795

INTERVENTIONS:
Drug: GSK1120212 (trametinib) — Trametinib dose is 1.5 mg orally once per day
  Other Names: Trametinib
Drug: GSK2141795 — The dose of GSK2141795 is 50 mg orally once per day

SUMMARY:
This research study is evaluating the combination of two drugs called GSK1120212 (trametinib) and GSK2141795 as a possible treatment for recurrent or persistent cervical cancer. Trametinib and GSK2141795 are drugs that may stop cancer cells from growing. Trametinib is a MEK inhibitor - it blocks a protein called MEK that is commonly overactive in tumor cells. GSK2141795 is an AKT inhibitor which blocks a pathway in cancer cells that is commonly overactive in tumor cells called the PI3kinase pathway. In this research study, the investigator is looking to see whether the combination of Trametinib and GSK2141795 is useful in treating recurrent and persistent cervical cancer.

Additionally, the investigator is looking to see if participants whose tumors contain a particular genetic make-up will have better response to combination trametinib and GSK2141795. Participants' tumors will be tested for mutations in genes which could make some cancers more susceptible to trametinib and GSK2141795.

DETAILED DESCRIPTION:
Before the research starts (screening): The participant will be asked to undergo some screening tests or procedures to find out if they can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that the participant does not take part in the research study. If the participant has had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about the participant's health, current medications, and any allergies.
* Physical exam, including height and weight
* An eye exam, by an eye specialist
* Performance status, the investigator will ask the participant questions about how they are able to carry on with your usual activities.
* Vital signs, including blood pressure, pulse, body temperature and respiratory rate
* An assessment of the participant's tumor by CT (Computerized Tomography) scan or MRI (Magnetic Resonance Imaging), of their chest, stomach area, and pelvis.
* Blood tests (approximately 2-3 tablespoons) including hematology, chemistry, liver function, kidney function, blood sugar levels, blood clotting levels
* Electrocardiogram (EKG), a test to check the participant's heart's rhythm
* Echocardiogram (ECHO), a test to check the participant's heart's structure and function.
* Serum pregnancy test if the participant are capable of becoming pregnant

If the results of the above tests show that the participant is eligible to participate in the research study, the participant will begin the study treatment. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.

If these tests show that the participant is eligible to participate in the research study, the participant will begin the study treatment. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.

Additional research procedures to be performed at the time of screening:

- Archival tumor testing: During this study, additional tests will be performed on a sample of the participant's original tumor that has been stored in your institution's tissue banks. These tests will be performed on tumor tissue samples from previous biopsies or surgeries for the participant's cancer. The research done on these samples will involve looking at DNA and proteins in the participant's cancer to see if researchers can learn more about the participant's type of cancer and understand how trametinib and GSK2141795 might work on their tumor. Testing of this sample will not require the participant to undergo any additional procedures.

TISSUE COLLECTIONS/OWNERSHIP: Participation in this protocol involves providing specimen(s) of the participant's tissue. Please know that if the investigator leaves the institution, the research and the tissue might remain at the DF/HCC or might be transferred to another institution.

* Additional Blood tests: Approximately 2 tablespoons of blood will be collected for research testing. This testing will involve looking at DNA and proteins in the participant's blood to compare them with those seen in their cancer. This will be drawn before the participant begin taking the study drug. These research sample collections are a required part of this research study. If the participant does not wish to undergo these procedures, the participant may not participate in this research study.
* Optional pre and post tumor biopsies: Before the participant begin receiving the study drug, your doctor will arrange for a procedure where your tumor will be biopsied. Your entire tumor or part of your tumor might be removed (excisional biopsy) or a small sample of the tumor might be removed using a needle (needle biopsy, fine needle aspirate) with guidance under radiographic studies. This will also occur before the participant begins treatment and between 2-4 weeks after treatment has started.

After the screening procedures confirm that the participant is eligible to participate in the research study:

Study Drugs:

If the participant decides to take part in this research study, the participant will be given a study drug diary for each treatment cycle. The participant will be asked to complete a drug diary to record when they took each dose or to give a reason if the participant did not take the study drugs. At the end of each cycle, the participant should return the pill bottles and all of the remaining pills prior to starting the next cycle. The participant will receive a new set of pills and new diary if the participant is to continue the next cycle.

Clinical Exams: During all cycles the participant will have a physical exam, and will be asked questions about their general health and specific questions about any problems that they might having and any medications the participant may be taking.

The participant can expect the following while they are a participant on this study.

At the beginning of each cycle (one cycle equals 28 days):

* Recording of any health problems, including side effects of the study drugs
* List of medications taken since the last visit
* Physical examination (including measurement of vital signs, such as blood pressure, breathing rate, heart rate, temperature and weight)
* Evaluation of the participant's performance status (the ability to carry on daily activities)
* Blood samples (approximately 2-3 tablespoons of blood will be taken) to evaluate the participant's blood counts, electrolytes, liver function, kidney function and blood sugar levels.
* EKG, a test to check the participant's heart's rhythm. This will be performed at the start on each cycle.

Once a week during the first cycle:

* The participant will be called by a member of the study team to record any health problems, including side effects from the study drugs and any changes in medications.
* Blood samples (approximately 1 teaspoon of blood will be taken) to evaluate their blood sugar levels. This can be done at a lab close to home. If the participant's doctor thinks that their blood sugars need further monitoring, the participant may have continued blood samples drawn to check their blood sugar weekly or daily past the first cycle.

Every 2 cycles:

* Blood samples (approximately 1 teaspoon of blood will be taken) to evaluate the participant's HgbA1C, a test that evaluates their blood sugar levels over a period of time. This can be done at a lab close to home.
* CT scan or MRI of your chest, stomach area, and pelvis to see if the participant's cancer is increasing, decreasing, or staying the same size. If the cancer is decreasing, the participant's doctor may schedule the participant for another CT scan in about one month to check it again.
* ECHO, a test to check the participant's heart's structure and function

At the end of the study:

* Recording of any health problems, including any side effects from the study drugs.
* List of medications taken since the last visit
* Physical examination (including measurement of the participant's vital signs, such as blood pressure, breathing rate, heart rate, temperature, and weight.)
* Evaluation of the participant's performance status (their ability to carry on daily activities).
* Blood samples (approximately 2-3 tablespoons of blood will be taken) to evaluate the participant's blood counts, electrolytes, liver function, kidney function, blood sugar level, and HgbA1C.

After the final dose of the study drug:

The investigator would like to keep track of the participant's medical condition for up to 3 years after the participant completes the study. The investigator would like to do this by calling the participant on the telephone or seeing the participant in clinic for evaluation of their status, disease and current therapy. Keeping in touch with the participant and checking their condition routinely helps us look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic cervical cancer of any histology
* Measurable disease by RECIST 1.1.
* Prior Therapy:
* At least one prior chemotherapy regimen for management of cervical cancer. Radiation-sensitizing chemotherapy will not be counted as a systemic chemotherapy regimen
* Patients can have received one additional regimen for treatment
* No prior receipt of PI3K or RAS-ERK pathway inhibitors
* Age ≥ 18 years
* Life expectancy > 3 mos
* ECOG performance status ≤ 2
* Participants must have normal organ function as defined below:
* Absolute Neutrophil Count (ANC)≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin > 9.0/dL
* AST (SGOT) and ALT (SGPT) ≤ 2.5 × institutional ULN
* Total Bilirubin within normal institutional limits
* Albumin ≥ 2.5 g/dL
* Creatinine ≤ upper limit of institutional normal or creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal or ≥ 50 mL/min 24-hour creatinine clearance
* Normal LVEF
* Normal fasting Blood Glucose
* Availability of a formalin fixed paraffin embedded (FFPE) block of cancer tissue
* Normal blood pressure (systolic < 140 mmHg and diastolic < 90 mmHg)
* Women of childbearing potential must agree to use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Toxicities of prior therapy (excepting alopecia) should be resolved to ≤ grade 1
* Ability to tolerate oral medications and no malabsorption
* Ability to sign an informed consent

Exclusion Criteria:

* No previous chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C,) or radiation therapy within 2 weeks prior to entering the study
* No use of investigational agents nor have participated in an investigational trial within the past 4 weeks (or five half-lives whichever is shorter; with a minimum of 14 days from the last dose).
* Presence of active GI disease that could affect GI absorption or predispose a subject to GI ulceration.
* Evidence of mucosal of internal bleeding
* Major surgery within the last 4 weeks
* No Type 1 diabetes; however, patients with Type 2 diabetes are eligible if diagnosed ≥ 6 months prior to enrollment and if hemoglobin A1C (HbA1C) ≤ 8% at screening.
* Symptomatic or unstable brain metastases or asymptomatic and untreated but > 1 cm in the longest dimension
* Symptomatic or untreated leptomeningeal or spinal cord compression.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: the following cancers are eligible if diagnosed and treated within the past 3 years: breast cancer in situ and basal cell or squamous cell carcinoma of the skin, stage I colon carcinoma confined to a polyp.
* Any serious and/or unstable pre-existing medical disorders
* Known infection with HIV, Hepatitis B Virus, or Hepatitis C Virus
* Chronic use of drugs that are strong inhibitors or inducers of p450 CYP3A4
* known immediate or delayed hypersensitivity reaction or idiosyncrasy to study drugs
* History of interstitial lung disease or pneumonitis.
* Presence of cardiac metastases
* Subject with intra-cardiac defibrillators or pacemaker.
* History or current evidence / risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* History of RVO or CSR, or predisposing factors to RVO or CSR
* Visible retinal pathology as assessed by ophthalmic exam
* History or evidence of cardiovascular risk including any of the following
* QTcF≥ 480 msec ( ≥ 500 msec for subject with bundle branch block)
* History or evidence of current clinically significant uncontrolled arrhythmias. (Exception: controlled atrial fibrillation for >30 days prior to randomization)
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months of study entry.
* Class II or higher congestive heart failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula A. Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Response Rate for the Combination of GSK1120212 (Trametinib) and GSK2141795 in Patients With Recurrent or Persistent Cervical Cancer.
Description: Response rate will be assessed by RECIST version 1.1.
Time Frame: 2 Years
Population: Response rate assessed by RECIST version 1.1.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Number analyzed (Participants) | 14
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 8
  Unevaluable | 2
  Progressive Disease | 3

2. Secondary Outcome: Duration of Progression-free (PFS)
Description: The duration of progression-free (PFS) following initiation of therapy with GSK1120212 (trametinib) and GSK2141795 will be measured.
Time Frame: 2 Years
Population: PFS events were determined by RECIST 1.1, clinical progression and death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Number analyzed (Participants) | 11
months | 3.7 [1.9 to NA] — Study was stopped prematurely, insufficient number of participants with events.

3. Secondary Outcome: Toxicity of GSK1120212 (Trametinib) and GSK2141795 as Measured by the Number of Participants With Adverse Events
Description: Toxicity was assessed for this combination by version 4.0 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) in this cohort of patients. Toxicities reported were deemed related to study treatment.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Number analyzed (Participants) | 14
Participants | 14

4. Secondary Outcome: Mutation and Co-mutation Rates of Genes in the PI3K and RAS ERK Signaling Pathways in Recurrent Cervical Cancer Using High Throughput Targeted Mutational Analysis on Participant Tumor Samples.
Description: The mutation and co-mutation rates of genes in the PI3K and RAS ERK signaling pathways in recurrent cervical cancer will be interrogated using high throughput targeted mutational analysis on participant tumor samples.
Time Frame: 2 Years
Population: Observed mutations and amplifications in genes related to PI3K or RAS signaling in the 13 patients with tissue available for testing. One patient did not have archival tissue available for testing, five patients did not have detected alterations.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Number analyzed (Participants) | 13
Participants
  Adenocarcinoma: number analyzed (Participants) | 5
  Adenocarcinoma: PIK3CA mutation | 2
  Adenocarcinoma: PIK3CA amplification | 1
  Adenocarcinoma: KRAS abberation | 2
  Squamous Cell Carcinoma: number analyzed (Participants) | 2
  Squamous Cell Carcinoma: PIK3CA mutation | 2
  Squamous Cell Carcinoma: PIK3CA amplification | 0
  Squamous Cell Carcinoma: KRAS abberation | 0
  Mucinous: number analyzed (Participants) | 1
  Mucinous: PIK3CA mutation | 0
  Mucinous: PIK3CA amplification | 0
  Mucinous: KRAS abberation | 1

5. Secondary Outcome: Overall Survival
Description: Overall survival will be determined for subjects on this study
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
Number analyzed (Participants) | 11
months | 14.8 [6.7 to NA] — Study stopped prematurely, insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Arm/Group | GSK1120212 (Trametinib) and GSK2141795
All-Cause Mortality (participants affected / at risk) | 8/14
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1120212 (Trametinib) and GSK2141795 (N=14)
Thromboembolic event (Blood and lymphatic system disorders) | 2 (2)
colonic perforation (Gastrointestinal disorders) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1)
Retinal pigment epithelial detachment (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1120212 (Trametinib) and GSK2141795 (N=14)
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT01958112/Prot_SAP_000.pdf